CLINICAL TRIAL: NCT07384559
Title: Exploratory Study Investigating the Urinary Bladder During Intermittent Catheterization in Healthy and Spinal Cord Injured Male and Female Subjects Using an Upright MRI Scanner
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP386
Record Dates: First submitted 2026-01-19; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Retention, Urinary
MeSH Terms: conditions — Urinary Retention | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: To obtain usable MRI 3D images of lower urinary tract and surroundings during voiding (healthy subjects) and during bladder emptying with IC (healthy subjects and SCI subjects).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI scan (Other): MRI scan of SCI and healthy male/female subjects during catheterization
  Interventions: Other: MRI scan

INTERVENTIONS:
Other: MRI scan — MRI scan of SCI and healthy male/female subjects during catheterization

SUMMARY:
This is an exploratory study investigating morphological and physiological changes of the lower urinary tract and surrounding structures during IC use in individuals with SCI, and during normal voiding and IC use in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Has given written informed consent
2. Is at least 18 years old
3. Has full legal capacity
4. Is able (assessed by investigator) and willing to adhere to study procedures during study duration
5. Is able (assessed by investigator) to remain seated in the MRI scanner for minimum 20 minutes*
6. Known with SCI for a minimum of 1 year*
7. Has used IC as primary bladder emptying method for at least 3 months* * Only for SCI subjects

Exclusion Criteria:

1. Is participating in any other clinical investigation during this investigation
2. Has previously completed this investigation
3. Has any known allergic or hypersensitive reactions to any device or its ingredients used in the investigation
4. Is pregnant
5. Has had surgical procedures performed in the lower urinary tract.
6. Has active/recurrent bladder cancer
7. Has experienced autonomic dysreflexia within the last 2 years
8. Has any MRI-scanning contraindications, according to MR check list provided by the site (e.g. active implants like pacemaker, cochlear implant, event recorder, implanted insulin pump)
9. Has symptoms of UTI at times of inclusion, as judged by the investigator.
10. Has a body weight that exceeds the maximum of 150kg max

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Is the quality of the 3D MRI images performed at Visit 2 sufficient for further use/analysis? (Y/N). | up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Walter Wigger-Alberti, M.D., Principal Investigator — Eurofins bioskin GmbH

IPD SHARING:
Plan to Share IPD: Undecided